CLINICAL TRIAL: NCT00991185
Title: CSF Pharmacokinetics of Antimicrobials in Children
Brief Title: Cerebrospinal Fluid (CSF) Pharmacokinetics of Antimicrobials in Children
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00013132; 5U10HD045962 (NIH)
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2024-04-15 (Actual); Status verified 2014-06

CONDITIONS: Infections
Keywords: Infections in Children
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — CSF, Blood, urine, bronchial, salivary, peritoneal, wound/abscess
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to learn more about antimicrobials, especially drug levels in the CSF that would normally be used in young children as part of standard care. These drugs are approved by the Food and Drug Administration (FDA) for treating infections. They are used extensively in children in the United States, but they have not been extensively studied in children or babies. The investigators do not have very much information on how children and babies handle these drugs; that is, how long it takes for the drugs to be removed from the blood circulation and to pass out of the body and how much goes into the central nervous system. The investigators also do not have good information to guide how often the investigators should give the drugs to children and babies to get the maximum effect on infections with the minimum amount of drug. Thus, the investigators will collect more information about how these drugs should be used in children and babies by doing this drug levels research study.

ELIGIBILITY:
Inclusion Criteria:

* Children receiving antimicrobial agents and having cerebrospinal fluid collected as part of standard of care

Exclusion Criteria:

* Lack of consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (<18) receiving antimicrobial agents and having cerebrospinal fluid collected as part of standard of care
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2009-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Autmizguine J, Moran C, Gonzalez D, Capparelli EV, Smith PB, Grant GA, Benjamin DK Jr, Cohen-Wolkowiez M, Watt KM. Vancomycin cerebrospinal fluid pharmacokinetics in children with cerebral ventricular shunt infections. Pediatr Infect Dis J. 2014 Oct;33(10):e270-2. doi: 10.1097/INF.0000000000000385. PMID 24776517

RESULTS

PARTICIPANT FLOW:
Groups:
- Vancomycin: children that received vancomycin per standard of care
Period: Overall Study
Arm/Group | Vancomycin
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vancomycin
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 4 [0.2 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: CSF:Serum Ratio of Vancomycin
Description: CSF:serum ration of vancomycin
Time Frame: within 1 week of drug administration
Measure: Median (Full Range); unit: ratio
Arm/Group | Vancomycin
Number analyzed (Participants) | 8
ratio | 0.08 [0 to 0.66]

ADVERSE EVENTS:
Arm/Group | Vancomycin
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No